CLINICAL TRIAL: NCT02496442
Title: Aqueduct Irrigation System Clinical Protocol: Medical Device Investigational Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Flowmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CIS-01
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Prostatic Hyperplasia; Kidney Calculi; Bladder Tumors
Keywords: Transurethral Resection of Prostate; Cystoscopy; PCNL; RERAS; Urethroscopy
MeSH Terms: conditions — Prostatic Hyperplasia; Kidney Calculi; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- using Aqueduct (Active Comparator): Patients passing procedures with Aqueduct
  Interventions: Device: Aqueduct
- Not using Aqueduct (No Intervention): Patients passing the standard procedures

INTERVENTIONS:
Device: Aqueduct — Using Aqueduct in procedures to continuously supply the irrigation solutions
  Arms: using Aqueduct

SUMMARY:
A. Synopsis

1. This protocol comes to direct the experiment to be performed on the Aqueduct Automatic Continuous Irrigation system.
2. The Aquaduct System is aimed at reducing risks to the patient by decreasing the irrigation fluid pressure he may be exposed to, reducing the procedure time and therefore the anesthesia time, reducing the manual handling of the sterile bags and the risk of contamination and more.
3. In general since there is no new procedure suggested and the equipment does not actually come into contact with the human body in any direct way, there is no need to have a clinical study for the regulation purpose. The reason for performing this experiment is to demonstrate the new system and to find out the best way to operate it in order to improve the process and reduce risks.
4. This information will serve the development of most suitable automation solution for achieving the long desired continuous irrigation.
5. The experiment will be performed in the OR in MIS procedures, and will replace the standard gravitational manual method of performing the irrigation. The surgeons and the medical staff of the OR will be directed with the set up and operation of the system prior to using it. The experiment will be accompanied at all times with a knowledgeable representative of the research originator.
6. A maximum of 30 procedures will be analyzed during a period of approximately one month. The surgeons and the medical staff will report their impression of using the system during the procedures and will recommend the best settings achieved.

This information will be used to improve the system performance and design.

DETAILED DESCRIPTION:
1.0 Purpose of the Investigation

1.1 Name of investigational device:

Aqueduct model CIS-01

1.2 Intended use of the investigational device:

Automatic Continuous Irrigation in Endoscopic procedures.

1.3 Objectives of the clinical investigation:

1.3.1 Primary objective.

Demonstrating the efficacy of the use of the Aqueduct system in:

* Continuity of flow
* Ease of operation

1.3.2 Secondary objective(s).

* Evaluation of potential safety issues associated with the use of the device;
* Evaluation of device design;
* Assessing certain human factors (e.g., patient or operator) associated with the use of the device; or
* Other specified device characteristic or device application consideration.

1.4 Anticipated duration of the clinical investigation:

1 Month

2.0 Clinical Protocol

2.1 Title of clinical protocol:

Operation of automatic irrigation controller in endoscopic procedures

2.1.1 Protocol number. Version 01

2.1.2 Version number and date. Version 1, March 4, 2015

2.2 Study design:

2.2.1 General study design.

During this study the system will be used by surgeons after teaching of the system capabilities, as they feel correct.

Surgeons will setup the system to supply solution flow with limiting pressure. Increase of flow during operation as they require limited by the set pressure and by safety valve to 180 cmH2O.

Following each procedure a case report form (attached in chapter 11 below) will be filled, reporting single experiment results.

Both cases using the system or standard procedures not using it will be reported and summarized in a table.

The results will serve to analyze the equipment performance and efficacy.

2.3 Subject selection:

2.3.1 General characteristics of the proposed subject population(s).

Regular endoscopic procedures patient(s).

There is no difference between standard procedure and using the Aqueduct. Only improvements without risks are expected.

2.3.2 Anticipated number of research subjects.

Up to 30 patients will be enrolled to the experiment. They will have to sign the consent form explaining the experiment

2.3.3 Inclusion criteria.

Any adult over the age of 18 who is candidate to endoscopic procedure is suitable for the experiment

2.3.4 Exclusion criteria.

Only adults over the age of 18.

2.4 Study procedures:

2.4.1 Screening procedures.

The surgeon performing the operation will suggest the use of the Aqueduct to relevant patients. He will explain the principles of the system the advantages and risks and their mitigation.

If patient agrees and will sign the consent form he will be enrolled.

2.4.2 Study treatment or diagnostic product procedures.

The study will include series of procedures in which the surgeons will utilize the Aqueduct for the irrigation instead of the use of the current bags pole.

The surgeons will inspect the parameters and settings of the Aqueduct, experiment any values that may ease the procedure.

In general they will try the minimal flow and minimal pressure to be used efficiently. If needed they will be able to increase or decrease the flow and the limiting pressure.

In subsequent procedures the surgeons will use the settings achieved in the previous procedures.

After 10 procedures we will collect the best settings for future default setup of the Aqueduct for each procedure.

2.4.3 Follow-up procedures.

2.4.3.1 Procedures to assess efficacy:

As the standard procedures calls for gravitational flow from 60 Cm above the patient, which creates free flow of between 350 to 270 milliliter per minute and nominal pressure which is above 60 cm H2O, the efficacy will be proved by the following:

1. Nominal flow below 300ml/min
2. Nominal pressure below 60cm H2O As lower the results will be lesser is the risk to the patient .

2.4.3.2 Procedures to assess safety:

Closing the input tap of the resectoscope will lead to operation of the pressure relief valve at 180 cm H2O showing the protection achieved from overpressure.

2.4.4 Schedule of activities (Study Table).

Incorporated as a referenced attachment is a table that summarizes the protocol procedures that will be performed at screening, for treatment or diagnosis, and at follow-up.

2.5 Study outcome evaluations:

2.5.1 Study endpoints.

After each procedure the surgeon will fill the protocol summary (per attachment in chapter 11 below): with his observations

1. If continuous flow was maintained during the procedure
2. If the ease of use of the equipment was acceptable
3. Any ideas for improvements in next system generations The study endpoint will be after at least 10 procedures using the Aqueduct.

The secondary objectives will be satisfied by the ideas for improvements in next system generations.

2.5.2 Sample size determination.

There is no need to perform any clinical trial. The justification for the sample size selected is just by the estimated time needed to evaluate the system.

2.5.3 Outcome data and data analysis.

Average of the observations and/or measurements that result from using the system efficiently will be the primary results of the experiment.

The, secondary results or outcomes of the clinical study are the suggestions for improvement.

The results will be used to reach a production model of the Aqueduct. 3.0 Risk Analysis

3.1 Anticipated risks:

Risks to patients are limited to the system extracting overpressure to the organs being operated.

The steps taken to reduce this risks are triple

1. Set up of the system is to lower parameters of pressure than the values used in current procedures
2. A pressure sensor is incorporated within the Y-Set providing the pressure readings and preventing overpressure.
3. In case of the system failure to control a low pressure a mechanical safety valve is set to 180 cm H2O and prevents any risk of larger pressure.
4. During the operation pressure reading appears on the screen and a warning message appears to the surgeon who can decide to stop the use of the Aqueduct and move to the standard procedure. The system is designed to ease of transferring the solution bags and the Y-Set to a standard gravitational activated pole.

   Since the overpressure is immediately detected and acted upon there is no real risk but just benefit to the patient.

   The benefit can be assessed by the % of flow from the average 330ml/min without the system and the % of pressure from the minimal 60 cmH2O used in the standard procedure.

   3.2 Adverse event recording/reporting

   3.2.1 Adverse event definitions.

   Adverse effect. Any untoward medical occurrence in a clinical study of an investigational device; regardless of the causal relationship of the problem with the device or, if applicable, other study treatment or diagnostic product(s).

   Associated with the investigational device or, if applicable, other study treatment or diagnostic product(s). There is a reasonable possibility that the adverse effect may have been caused by the investigational device or, if applicable, the other study treatment or diagnostic product(s).

   Disability. A substantial disruption of a person's ability to conduct normal life functions.

   Life-threatening adverse effect. Any adverse effect that places the subject, in the view of the investigator-sponsor, at immediate risk of death from the effect as it occurred (i.e., does not include an adverse effect that, had it actually occurred in a more severe form, might have caused death).

   Serious adverse effect. Any adverse effect that results in any of the following outcomes: death, a life-threatening adverse effect, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
   * Hospitalization shall include any initial admission (even if less than 24 hours) to a healthcare facility as a result of a precipitating clinical adverse effect; to include transfer within the hospital to an intensive care unit. Hospitalization or prolongation of hospitalization in the absence of a precipitating, clinical adverse effect (e.g., for a preexisting condition not associated with a new adverse effect or with a worsening of the preexisting condition; admission for a protocol-specified procedure) is not, in itself, a serious adverse effect.

   Unexpected adverse effect. Any adverse effect, the frequency, specificity or severity of which is not consistent with the risk information described in the clinical study protocol(s) or elsewhere in the current IDE application, as amended.

   Unanticipated adverse device effect. Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or IDE application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

   3.2.2 Eliciting adverse effect information.

   Clinical study subjects will be routinely questioned about adverse effects at study visits.

   3.2.3 Recording and assessment of adverse effects.

   All observed or volunteered adverse effects (serious or non-serious) and abnormal test findings, regardless of treatment group, if applicable, or suspected causal relationship to the investigational device or, if applicable, other study treatment or diagnostic product(s) will be recorded in the subjects' case histories. For all adverse effects, sufficient information will be pursued and/or obtained so as to permit 1) an adequate determination of the outcome of the effect (i.e., whether the effect should be classified as a serious adverse effect) and; 2) an assessment of the casual relationship between the adverse effect and the investigational device or, if applicable, the other study treatment or diagnostic product(s).

   Adverse effects or abnormal test findings felt to be associated with the investigational device or, if applicable, other study treatment or diagnostic product(s) will be followed until the effect (or its sequelae) or the abnormal test finding resolves or stabilizes at a level acceptable to the investigator-sponsor.

   3.2.3.1 Abnormal test findings:

   An abnormal test finding will be classified as an adverse effect if one or more of the following criteria are met:

   • The test finding is accompanied by clinical symptoms.
   * The test finding necessitates additional diagnostic evaluation(s) or medical/surgical intervention; including significant additional concomitant drug or other therapy. (Note: simply repeating a test finding, in the absence of any of the other listed criteria, does not constitute an adverse effect.)
   * The test finding leads to a change in study dosing or exposure or discontinuation of subject participation in the clinical study.
   * The test finding is considered an adverse effect by the investigator-sponsor.

   3.2.3.2 Causality and severity assessment:

   The investigator-sponsor will promptly review documented adverse effects and abnormal test findings to determine 1) if the abnormal test finding should be classified as an adverse effect; 2) if there is a reasonable possibility that the adverse effect was caused by the investigational device or, if applicable, other study treatment or diagnostic product(s); and 3) if the adverse effect meets the criteria for a serious adverse effect.

   If the investigator-sponsor's final determination of causality is "unknown and of questionable relationship to the investigational device or, if applicable, other study treatment or diagnostic product(s)", the adverse effect will be classified as associated with the use of the investigational device or study treatment or diagnostic drug product(s) for reporting purposes. If the investigator-sponsor's final determination of causality is "unknown but not related to the investigational device or, if applicable, other study treatment or diagnostic product(s)", this determination and the rationale for the determination will be documented in the respective subject's case history.

   3.2.4 Reporting of adverse effects to the FDA. )

   The investigator-sponsor will submit a completed Form FDA 3500 A to the FDA's Center for Devices and Radiological Health for any observed or volunteered adverse effect that is determined to be an unanticipated adverse device effect. A copy of this completed form will be provided to all participating sub-investigators.

   The completed Form FDA 3500 A will be submitted to the FDA as soon as possible and, in no event, later than 10 working days after the investigator-sponsor first receives notice of the adverse effect.

   If the results of the sponsor-investigator's follow-up evaluation show that an adverse effect that was initially determined to not constitute an unanticipated adverse device effect does, in fact, meet the requirements for reporting; the investigator-sponsor will submit a completed Form FDA 3500 A as soon as possible, but in no event later than 10 working days, after the determination was made.

   For each submitted Form FDA 3500 A, the sponsor-investigator will identify all previously submitted reports that that addressed a similar adverse effect experience and will provide an analysis of the significance of newly reported adverse effect in light of the previous, similar report(s).

   Subsequent to the initial submission of a completed Form FDA 3500 A, the investigator-sponsor will submit additional information concerning the reported adverse effect as requested by the FDA.

   3.2.5 Reporting of adverse effects to the responsible IRB.

   In accordance with applicable policies of the medical centre Institutional Review Board (IRB), the investigator-sponsor will report, to the IRB, any observed or volunteered adverse effect that is determined to meet all of the following criteria: 1) associated with the investigational device or, if applicable, other study treatment or diagnostic product(s); 2) a serious adverse effect; and 3) an unexpected adverse effect. Adverse event reports will be submitted to the IRB in accordance with the respective IRB procedures.

   Applicable adverse effects will be reported to the IRB as soon as possible and, in no event, later than 10 calendar days following the investigator-sponsor's receipt of the respective information. Adverse effects which are 1) associated with the investigational drug or, if applicable, other study treatment or diagnostic product(s); 2) fatal or life-threatening; and 3) unexpected will be reported to the IRB within 24 hours of the investigator-sponsor's receipt of the respective information.

   Follow-up information to reported adverse effects will be submitted to the IRB as soon as the relevant information is available. If the results of the sponsor-investigator's follow-up investigation show that an adverse effect that was initially determined to not require reporting to the IRB does, in fact, meet the requirements for reporting; the investigator-sponsor will report the adverse effect to the IRB as soon as possible, but in no event later than 10 calendar days, after the determination was made.

   3.3 Withdrawal of subjects due to adverse effects:

   In any case that the researcher decides that the subject is unsuitable for the experiment the subject will be withdrawn from the study.

   There will be no replacement and the endpoint may include less than planned subjects.

   4.0 Description of the Investigational Device

   The robotic technology is based on using the same solution bags. This electro-mechanic system will replace the manual bag-switching procedure with an automatic one.

   The system consists of several-sub mechanisms that identify when the bag solution is about to end, opens a flow from a buffer bag, pulls the spike of the Y-set from the empty bag, moves the spike to a new bag, removes its protective cover, spikes it and switches the flow from the buffer bag to the current bag - thus enabling a continuous irrigation. The system builds flow and pressure according to the procedure needs and enables the surgeon for the first time, to directly control it by a switch or a foot pedal allowing him to clear the visibility of the surgical site whenever it drops, as often happens during surgery due to excessive bleeding..

   The problems we solve:

1. Stoppage of fluid flow (no timely fluid bag replacement by nurse) 2. Physician control of the flow to prevent vision block by excess bleeding 3. Prolonged operation time 4 Glycinemia risk to the patient 5. Urethra injuries when entering the endoscope 6. Post operation blood clots The design was created to ensure a "user-friendly fool-proof " system. Flow Med offers for purchase the electro-mechanic system along with the disposable Y-sets designed exclusively for the Flow Med system

A microcontroller is supervising the operation of the system and sets the correct control algorithm to provide continuous flow.

2 Heads are incorporated. One in a fixed position and one rotating under the hanging bags on the carousel. Each of the heads include 3 stepper motors one to remove the caps of the bags, one to move the spike in and ut of the bag and one to open or close the flow.

A peristaltic pump is used to create the required flow.

The following sensors are included in the system:

1. Weight sensor - measuring the weight of the bags helping to decide on the time to switch bags
2. Pressure sensor in the system main body with a sterile pressure capin the Y-Set helping to prevent overpressure

A Safety relief valve at 180 cmH2O is incorporated in the Y-Set to prevent overpressure.

A safety switch prevents movement of the motors when the front door is opened.

The covers are secured with screws to prevent their removal.

5.0 Monitoring Procedures

The sponsor-investigator will permit direct access to the study monitors and appropriate regulatory authorities to the study data and to the corresponding source data and documents to verify the accuracy of these data.

The system was designed according to ISO14385 standard. Electrical safety testing has been performed to IEC 60601-1 and Electromagnetic Compatibility (EMC) testing has been tested according to IEC 60601-1-2 in ITL (Israel Test Laboratories) and has their certificate to show it passed the standards tests.

Appendix:

1. Case Report Form - reporting standard procedure results

Date:_________ Place:_________ Procedure type:______________ Number of bags used: _________________ Procedure time:_______________ Height of bags above patient:_____________ Times extra pressure applied to the bags:_________

Observations on flow continuity during the procedure:

1. Was continuous flow maintained during the procedure?
2. Would the offered system ease the procedure?
3. Any ideas for improvements in next system generations ____________________________________________________________________________________________________________________________

Other difficulties during the procedure:

______________________________________________________________

______________________________________________________________

Name:__________ Signature:__________

2. Case Report Form - reporting single experiment results

Date:_________ Place:_________ Procedure type:______________ Number of bags hanged before starting: ______

Changes in parameters set up prior to starting:

____________________________________________

Changes for optimal parameters after the experiment:

______________________________________________

Description of the operation during the procedure:

Parameter Value Procedure Time Bags used Foot pedal used Number of times foot pedal operated Number of steps used each time Closing the surgeons input tap result Closing the surgeon exit tap result Pressure protection performance Nominal Flow Nominal Pressure Maximal flow Maximal Pressure Min operating Flow Min operating Pressure Difficulties

Suggestions

Researcher name Researcher signature

1. Was continuous flow maintained during the procedure?
2. Is the ease of use of the equipment acceptable?
3. Any ideas for improvements in next system generations

ELIGIBILITY:
Inclusion Criteria:

* All patients passing the specific procedures set on the Aqueduct

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
continuous flow was maintained during the procedure | 3 Months
  evaluation of the continuous nature of the treatment using the Aqueduct
Ease of use | 3 months
  get qualitative assesment of the ease compared to standard procedure

SECONDARY OUTCOMES:
ideas for improvements | 3 Months
  ideas for improvements in next system generations.

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Moskovitz, Prof., Principal Investigator — Bnei-Zion

REFERENCES:
- [Background] i.